CLINICAL TRIAL: NCT02978170
Title: A New Guide for Our Guided-Bronchoscopy: The Use of Cone-Beam CT to Enhance Navigation and Diagnostic Yield of RP-EBUS and Hybrid Bronchoscope for Peripheral Lung Nodules Suspicious for Malignancy: A Pilot Study
Brief Title: CBCT in Guiding Bronchoscopy in Patients With Lung Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-0466; NCI-2017-00628 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0466 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Pulmonary Mass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (CBCT) (Experimental): Patients undergo CBCT during standard of care bronchoscopy.
  Interventions: Procedure: Cone-Beam Computed Tomography

INTERVENTIONS:
Procedure: Cone-Beam Computed Tomography — Undergo CBCT

SUMMARY:
This pilot clinical trial studies how well cone-beam computed tomography (CBCT) works in guiding bronchoscopy in patients with lung lesions. CBCT during bronchoscopy may help doctors to biopsy lung lesions that are harder to reach.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe the feasibility of using CBCT as an additional aid to guided-bronchoscopy with radial probe endobronchial ultrasound (RP-EBUS)/hybrid scope for the diagnosis of peripheral lung nodules.

SECONDARY OBJECTIVES:

I. Describe the proportion of patients with peripheral nodules undergoing bronchoscopy in whom the lesion is identified by RP-EBUS (RP-EBUS-navigation yield) and confirmed with CBCT.

II. Describe the proportion of patients with peripheral nodules undergoing bronchoscopy in whom the lesion is identified by RP-EBUS and samples are diagnostic (diagnostic yield-RP-EBUS).

III. Describe the proportion of patients with peripheral nodules undergoing bronchoscopy in whom the lesion is identified by RP-EBUS, samples were non-diagnostic, and CBCT prompted further tool re-location (i.e. change of needle angle, change of tool) leading to diagnosis.

IV. Describe the proportion of patients with peripheral nodules undergoing bronchoscopy in whom the lesion is not identified by RP-EBUS, and CBCT-aided navigation allowed the operator to reach the lesion (CBCT-added navigation yield).

V. Describe the proportion of patients with peripheral nodules undergoing bronchoscopy in whom the lesion is not identified by RP-EBUS and CBCT-aided navigation allowed the operator to reach the lesion and obtain a diagnosis (CBCT-added diagnostic yield).

VI. Describe the relationship between RP-PROBE and target (contact/no contact; central/peripheral).

VII. Describe the relationship between needle tip and target (contact/no contact; central/peripheral).

VIII. Describe the influence of points 6 and 7 on diagnostic yield. IX. Describe fluoroscopy time. X. Describe estimated amount of radiation generated by CBCT use. XI. Describe bronchoscopy time (first scope in/last scope out). XII. Describe the proportion of patients in whom molecular analysis for lung cancer (i.e. EGFR, K-RAS, ALK) can be performed.

OUTLINE:

Patients undergo CBCT during standard of care bronchoscopy.

After completion of study, patients with lesions found not to be cancerous are followed up for 6 months to watch for changes (standard care).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing guided-bronchoscopy for diagnosis of peripheral lung lesion/s > 1 and < 3 cm in diameter located in the outer 2/3 of the lung fields

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patient with indications for mediastinal lymph node (LN) sampling per 13th American College of Clinical Pharmacy (ACCP) guidelines
* Patient with metastatic disease (from primaries other than lung) who have suspicious mediastinal or hilar LN that require sampling
* Patients with contraindication/s for general anesthesia (e.g., severe and active coronary artery disease, chronic obstructive pulmonary disease [COPD] with forced expiratory volume in 1 second [FEV1] < 1 liter, uncontrolled hypertension, increased intracranial pressure, history of intolerance to general anesthesia)
* Dementia or other severe cognitive impairment causing inability to understand or consent to the procedure and study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2019-05-04 (Actual); Study Completion 2019-05-04 (Actual)

PRIMARY OUTCOMES:
Feasibility based on percentage of patients where researchers can locate target and bronchoscopic tools with cone-beam computed tomography | Up to 6 months
  Will be considered feasible if researchers can locate target and bronchoscopic tools with cone-beam computed tomography in at least 80% of the patients (16 out of the 20 participants) that are enrolled.

SECONDARY OUTCOMES:
Proportion of patients with peripheral nodules undergoing bronchoscopy in different subsample | Up to 6 months
  Will conduct extensive descriptive analyses of the data collected. Descriptive statistics (e.g., frequencies, ranges, means, proportions, standard deviations, and measures of skewness and kurtosis), including 90% confidence intervals will be calculated. Will closely examine distribution characteristics of the variables using box plots, histograms, and scatter plots, where appropriate.
Localization of the tip with respect to targets | Up to 6 months
  Will assess the relationship between radial probe/needle tip and target. Will conduct extensive descriptive analyses of the data collected. Descriptive statistics (e.g., frequencies, ranges, means, proportions, standard deviations, and measures of skewness and kurtosis), including 90% confidence intervals will be calculated. Will closely examine distribution characteristics of the variables using box plots, histograms, and scatter plots, where appropriate.
Diagnostic yield | Up to 6 months
  Will assess the influence of points 6 and 7 on diagnostic yield. Descriptive statistics (e.g., frequencies, ranges, means, proportions, standard deviations, and measures of skewness and kurtosis), including 90% confidence intervals will be calculated. Will closely examine distribution characteristics of the variables using box plots, histograms, and scatter plots, where appropriate.
Amount of radiation generated by cone-beam computed tomography use | Up to 6 months
  Descriptive statistics (e.g., frequencies, ranges, means, proportions, standard deviations, and measures of skewness and kurtosis), including 90% confidence intervals will be calculated. Will closely examine distribution characteristics of the variables using box plots, histograms, and scatter plots, where appropriate.
Fluoroscopy/bronchoscopy time | Up to 6 months
  Descriptive statistics (e.g., frequencies, ranges, means, proportions, standard deviations, and measures of skewness and kurtosis), including 90% confidence intervals will be calculated. Will closely examine distribution characteristics of the variables using box plots, histograms, and scatter plots, where appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Casal, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Casal RF, Sarkiss M, Jones AK, Stewart J, Tam A, Grosu HB, Ost DE, Jimenez CA, Eapen GA. Cone beam computed tomography-guided thin/ultrathin bronchoscopy for diagnosis of peripheral lung nodules: a prospective pilot study. J Thorac Dis. 2018 Dec;10(12):6950-6959. doi: 10.21037/jtd.2018.11.21. PMID 30746241
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org